CLINICAL TRIAL: NCT06032351
Title: Construction and Validation of Dementia Care Management Competency: From Curriculum Integration to Outcome Evaluation
Brief Title: Construction and Validation of Dementia Care Management Competency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Huei-Ling Huang, Associate Professor, PhD, RN, Department of Gerontology and Health Care Management, College of Nursing, Chang Gung University of Science and Technology, Taoyuan, Taiwan, R.O.C, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NSTC 112-2410-H-255 -006 -MY2; NMRPF3N0081 (Other: Chang Gung University of Science and Technology)
Record Dates: First submitted 2023-08-21; First posted 2023-09-13 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Dementia
Keywords: Teaching Method; Medical Practice Management; Competence; Competency-Based Education
MeSH Terms: conditions — Dementia | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional teaching group (Other): conventional teaching methods
  Interventions: Other: Traditional classroom teaching course programs
- curriculum integration Group (Experimental): The curriculum integration group will receive two intervention phases, including an innovation-integrated curriculum for dementia care and an innovation-integrated curriculum for care management with Entrustable Professional Activities (EPAs) to guide learning and assessment of competency performance to equip students with dementia care management competency.
  Interventions: Other: Innovation-integrated curriculum for dementia care and care management

INTERVENTIONS:
Other: Innovation-integrated curriculum for dementia care and care management — The curriculum integration group will receive two intervention phases, including an innovation-integrated curriculum for dementia care and an innovation-integrated curriculum for care management with Entrustable Professional Activities (EPAs), lectures, Situated Simulation Learning, Team-based learning, and Objective Structured Clinical Examination(OSCE).
  Other Names: experimental group
  Arms: curriculum integration Group
Other: Traditional classroom teaching course programs — The conventional teaching group will receive only traditional classroom teaching course programs.
  Other Names: Control Group
  Arms: conventional teaching group

SUMMARY:
This study will use the concept of competency-based education to develop an innovative integrated curriculum with EPAs to guide learning and assessment of competency performance to equip students with dementia care management competency and cultivate professionals to meet the social trends and practical needs.

DETAILED DESCRIPTION:
This study will use the concept of competency-based education to develop an innovative integrated curriculum with EPAs to guide learning and assessment of competency performance to equip students with dementia care management competency and cultivate professionals to meet the social trends and practical needs. The first year is a preparation period for the development of the project, which focuses on developing research tools and teacher empowerment, and evaluating the effectiveness of the control group in implementing conventional teaching methods. The second year is the program testing, implementation and evaluation period, in which two phases of the intervention is conducted and the post-intervention phase of competency is evaluated. This study is expected to establish a competency-based innovative and integrated curriculum for dementia care management over a two-year period. The results of the study will be used as a reference for schools or practices in the development of competency-based curriculum integration.

ELIGIBILITY:
Inclusion Criteria:

* (1)Be at least 20 years old.

  (2)The students are freshmen majoring in the Department of Gerontology and Health Care Management, and taking the course on Dementia care.

  (3)Before taking the course on Dementia care, have taken courses on basic geriatric nursing.

  (4)voluntary participation

Exclusion Criteria:

* The students who suspension of schooling.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Demographic data of student | The investigators will collect demographic data of students on the day before the start date of the intervention.
  Include age, gender, education level, areas of studying, etc.
Dementia Care Professional Competency Assessment Scale | T0(Baseline), T1(Immediately after the intervention), T2(3 months after the intervention).
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 106-2511-S-255-002-MY3). The scale is used to evaluate dementia care competency in students (Huang et al., 2018).
  2. This Scale contains nine subscales (74 items), using Likert 5-point Likert scale from 1 to 5. A higher score means better competencies.
  3. This scale is used to evaluate the competence of students.
Problem solving, Teamwork Competency Assessment Scale | T0(Baseline), T1(Immediately after the intervention), T2(3 months after the intervention).
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 106-2511-S-255-002-MY3). There are 22 questions on this scale. The scale is used to evaluate the problem-solving and teamwork competency of students. (Huang et al. 2018).
  2. This scale contains 22 items.10 items were used to evaluate problem-solving competencies, 12 items were used to evaluate teamwork competencies. A higher score means better competencies.
  3. This scale is used to evaluate the competence of students. Change from Baseline problem-solving and teamwork competency at the end of the semester, and after students finish the clinical practice course.
Learning Satisfaction Scale | Immediately after the intervention.
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 106-2511-S-255-002-MY3). There are 9 questions on this scale. The scale is used to evaluate the learning satisfaction of students. (Huang et al. 2018).
  2. This Scale contains 9 items, using Likert 5-point Likert scale from 1 to 5. A higher score means high learning satisfaction.
  3. This scale is used to evaluate the learning satisfaction of students.
Performance in a summative OSCE test (OSCE scores) | Immediately after the intervention.
  1. Conduct Objective Structured Clinical Examination
  2. After the intervention, the study sample participated in the final OSCE exam. Their scores were compared. The minimum value was 0 while the maximum value was 100. The higher the score the better students had performed.
Qualitative interview | The investigators will conduct qualitative interviews using focus groups 3 months after the intervention.
  Conduct qualitative interviews with the curriculum integration group students, focusing on the effectiveness of the curriculum integration.

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Ling Huang, PhD, Study Chair — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Taiwan